CLINICAL TRIAL: NCT03656185
Title: Retrospective Chart Analysis of Elbow Arthroscopy for the Treatment of Osteoarthritis, Radiocapitellar Plica, Lateral Epicondylitis or Osteochondritis Dissecans
Brief Title: Elbow Arthroscopy Data Analysis
Acronym: EA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Orthopaedic Research & Innovation Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: ORIF.009
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Osteoarthritis Elbow Left; Osteoarthritis Elbow Right; Lateral Epicondylitis, Left Elbow; Lateral Epicondylitis, Right Elbow; Plica Syndromes; Osteochondritis Dissecans
MeSH Terms: conditions — Tennis Elbow; Synovitis; Osteochondritis Dissecans

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to evaluate preoperative objective measurements and operative objective measurements to determine if there is any effect to postoperative outcomes. Patients who were 13 years old or greater at the time of arthroscopic osteocapsular release were followed clinically and radiographically to determine best practice and optimal treatment and technique, risk and rate of complication, and postoperative outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. >13 years of age
3. Patients treated with elbow arthroscopy for elbow arthritis, radiocapitellar plica, osteochondritis dissecans or lateral epicondylitis.

Exclusion Criteria:

1. Non-English speaking
2. <13 years of age

Age Groups: Child, Adult, Older Adult
Study Population: All eligible patients of the principal investigator receiving elbow arthroscopy for any indication at St. Elizabeth Healthcare between January 1, 2010 and October 31, 2017 will be evaluated and included in the data analysis. We anticipate approximately 150 patients to be included in the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-03-15 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Patient Outcomes | preoperative to up to 8 years postoperative
  The Quick Disabilities of the Arm, Shoulder and Hand Score. Scale of 0-100, 100 being the best possible score
Patient Satisfaction: one question assessment | 2 years to 8 years postoperative
  one question assessment of the patients overall long term satisfaction with the outcome of the treatment.
Patient Outcomes | preoperative to up to 8 years postoperative
  Visual Analogue pain Scale. Scale is 0-10, 0 is no pain, 10 is the most pain

CONTACTS AND LOCATIONS:
Locations (1):
- The Orthopaedic Research & Innovation Foundation, Edgewood, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Undecided